CLINICAL TRIAL: NCT03511729
Title: Tau/P-Tau as Biomarkers of Anesthesia/Surgery-associated Neurocognitive Outcomes in Children
Brief Title: Tau/P-Tau and Neurocognitive Outcomes in Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Zhongcong Xie, Professor of Anesthesia, Massachusetts General Hospital
Other Study IDs: 2019P000757; 5R21HD098754-02 (NIH)
Record Dates: First submitted 2018-04-11; First posted 2018-04-30 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: General Anesthetics Toxicity; Postoperative Cognitive Dysfunction; Child Development
Keywords: Tau/P-Tau; biomarker; neurocognitive; outcomes; children
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The investigators will harvest 300ul blood of participants before and 3, 6 hours after the surgery. Urine, feces and saliva from these participants will also be harvested.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- A single exposure to general anesthesia: Participants who have surgery under general anesthesia (without anesthesia/surgery before)
- Multiple exposures to general anesthesia: Participants who have surgery under general anesthesia (had anesthesia/surgery before)

SUMMARY:
The proposed studies are aimed to measure Tau and P-Tau levels in pre- and postoperative blood, urine, feces and saliva, as well as to assess pre- and postoperative neurocognitive function in children (3 to 5 years old) who will have surgery under general anesthesia (single versus multiple exposures). The studies will establish a system to study biomarkers of the anesthesia/surgery-associated neurocognitive impairment in children and generate hypothesis that Tau or P-Tau serves as the biomarker of such neurocognitive impairment in children.

DETAILED DESCRIPTION:
This proposed studies have two specific aims:

1. To investigate the relationship between pre-operative or postoperative blood levels of Tau or P-Tau and neurocognitive outcomes. The working hypothesis is that pre- and postoperative blood Tau/P-Tau levels are higher in participants who develop neurocognitive impairment than those in the participants who do not develop it. The investigators will perform neurocognitive test before the surgery and then at 12 months after the surgery. The investigators will collect pre-operative and postoperative blood and measure Tau/P-Tau levels in the blood. Finally, the association of the changes in the Tau/P-Tau levels and neurocognitive scores will be assessed. More importantly, this Aim will establish an eligible: recruit ratio, retention rates, safety of the protocol, and power calculation, which will provide crucial information to guide better design of future R01 study.
2. To perform the feasibility studies of measuring Tau or P-Tau in urine, feces and saliva of the participants. The working hypothesis is that Tau/P-Tau in urine, feces or saliva of children can be measured. The investigators will use the nanobeam to measure Tau/P-Tau levels before and after the surgery. The investigators will then determine whether urine, feces and saliva can be used for the future studies to develop Tau/P-Tau as the biomarker of anesthesia/surgery-associated neurocognitive impairment in children.

ELIGIBILITY:
Inclusion Criteria:

1. between age 3 and 5 at the time of the first neurocognitive test;
2. scheduled for surgery under general anesthesia

Exclusion Criteria:

1. gestational age less than 36 weeks;
2. congenital heart disease that has required surgery or will require surgery or that requires ongoing pharmacotherapy;
3. known chromosomal abnormality or any other known acquired or congenital abnormalities which are likely to affect neurodevelopment;
4. known neurological injury such as cystic periventricular leukomalacia or grade 3 or 4 intra-ventricular hemorrhage (+/- post hemorrhage ventricular dilatation);
5. children for whom follow-up would be difficult for geographic or psychosocial reasons;
6. non-native English speaker (both child and parents);
7. severe visual or auditory disorder.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The investigators will enroll participants between age 3 and 5 years old who are scheduled for the surgery under general anesthesia from Shriners Hospital for Children or Boston Children Hospital.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Tau/P-Tau level before the surgery (baseline) | Before the surgery
  300 ul venous blood before the surgery will be collected from the inserted intravenous catheter to measure the levels of Tau/P-Tau
Blood Tau/P-Tau level at postoperative 3 hours | At 3 hours after the surgery
  300 ul venous blood at 3 hours after the surgery will be collected from the inserted intravenous catheter to measure the levels of Tau/P-Tau
Blood Tau/P-Tau level at postoperative 6 hours | At 6 hours after the surgery
  300 ul venous blood at 6 hours after the surgery will be collected from the inserted intravenous catheter to measure the levels of Tau/P-Tau

SECONDARY OUTCOMES:
Neurocognitive function before the surgery (baseline) | Before the surgery
  Cognitive function will be assessed by using a battery of neurocognitive tests before the surgery
Neurocognitive function at postoperative one year | At postoperative one year
  Cognitive function will be assessed by using a battery of neurocognitive tests at postoperative one year
Feces Tau/P-Tau level before the surgery (baseline) | Before the surgery
  Feces will be collected to measure the level of Tau/P-Tau before the surgery
Feces Tau/P-Tau level at postoperative one day | At postoperative one day
  Feces will be collected to measure the level of Tau/P-Tau at postoperative one day
Urine Tau/P-Tau level before the surgery (baseline) | Before the surgery
  Urine will be collected to measure the level of Tau/P-Tau before the surgery
Urine Tau/P-Tau level at postoperative one day | At postoperative one day
  Urine will be collected to measure the level of Tau/P-Tau at postoperative one day
Saliva Tau/P-Tau level before the surgery (baseline) | Before the surgery
  Saliva will be collected to measure the level of Tau/P-Tau before the surgery
Saliva Tau/P-Tau level at postoperative one day | At postoperative one day
  Saliva will be collected to measure the level of Tau/P-Tau at postoperative one day

CONTACTS AND LOCATIONS:
Overall Officials: Zhongcong Xie, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Boston Childrens Hospital, Boston, Massachusetts
  - Zhongcong Xie, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication will be available to other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data will be available 6 months after publication
Access Criteria: Principle investigator will review the requests and determine what information should be shared.
URL: https://clinicaltrials.gov/

REFERENCES:
- [Background] Wilder RT, Flick RP, Sprung J, Katusic SK, Barbaresi WJ, Mickelson C, Gleich SJ, Schroeder DR, Weaver AL, Warner DO. Early exposure to anesthesia and learning disabilities in a population-based birth cohort. Anesthesiology. 2009 Apr;110(4):796-804. doi: 10.1097/01.anes.0000344728.34332.5d. PMID 19293700
- [Background] Flick RP, Katusic SK, Colligan RC, Wilder RT, Voigt RG, Olson MD, Sprung J, Weaver AL, Schroeder DR, Warner DO. Cognitive and behavioral outcomes after early exposure to anesthesia and surgery. Pediatrics. 2011 Nov;128(5):e1053-61. doi: 10.1542/peds.2011-0351. Epub 2011 Oct 3. PMID 21969289
- [Background] Kalkman CJ, Peelen L, Moons KG, Veenhuizen M, Bruens M, Sinnema G, de Jong TP. Behavior and development in children and age at the time of first anesthetic exposure. Anesthesiology. 2009 Apr;110(4):805-12. doi: 10.1097/ALN.0b013e31819c7124. PMID 19293699
- [Background] Sun L. Early childhood general anaesthesia exposure and neurocognitive development. Br J Anaesth. 2010 Dec;105 Suppl 1(Suppl 1):i61-8. doi: 10.1093/bja/aeq302. PMID 21148656
- [Background] Ing CH, DiMaggio CJ, Whitehouse AJ, Hegarty MK, Sun M, von Ungern-Sternberg BS, Davidson AJ, Wall MM, Li G, Sun LS. Neurodevelopmental outcomes after initial childhood anesthetic exposure between ages 3 and 10 years. J Neurosurg Anesthesiol. 2014 Oct;26(4):377-86. doi: 10.1097/ANA.0000000000000121. PMID 25144506